CLINICAL TRIAL: NCT04421846
Title: COLETTE : Study of the Pathophysiology of Status Epilepticus and Dysimmune Encephalitis and Identification of Valuable Biomarkers
Brief Title: Study of Pathophysiology of Status Epilepticus and Dysimmune Encephalitis
Acronym: COLETTE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: APHP200306; 2020-A00053-36 (Other: ANSM)
Record Dates: First submitted 2020-06-04; First posted 2020-06-09 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Status Epilepticus; Dysimmune Encephalopathy
Keywords: Epilepsy; Status Epilepticus; Autoimmunity
MeSH Terms: conditions — Status Epilepticus; Epilepsy; Autoimmune Diseases | interventions — Blood Specimen Collection; Sodium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 : Status epilepticus (Other)
  Interventions: Other: Blood sampling, cerebrospinal fluid, stool sampling post-mortem cerebral tissues (NA for the Group 3)
- Group 2 : Dysimmune encephalitis (Other)
  Interventions: Other: Blood sampling, cerebrospinal fluid , post-mortem cerebral tissues (NA for the Group 3)
- Group 3 : Control patients (Other)
  Interventions: Other: Blood sampling, cerebrospinal fluid , post-mortem cerebral tissues (NA for the Group 3)

INTERVENTIONS:
Other: Blood sampling, cerebrospinal fluid , post-mortem cerebral tissues (NA for the Group 3) — Collection of biological samples and clinical/paraclinical data
  Arms: Group 2 : Dysimmune encephalitis; Group 3 : Control patients
Other: Blood sampling, cerebrospinal fluid, stool sampling post-mortem cerebral tissues (NA for the Group 3) — Collection of biological samples and clinical/paraclinical data
  Arms: Group 1 : Status epilepticus

SUMMARY:
COLETTE is an interventional study for which blood, cerebrospinal fluid and post-mortem tissues are collected in patients with status epilepticus or epilepsy associated to dysimmune encephalitis as well as in control patients, to better understand the pathophysiology of these severe epileptic disorders.

DETAILED DESCRIPTION:
Epilepsy is one of the most common neurological condition which concerns around 50 million people worldwide. Epilepsy is characterized by a lasting predisposition to generate seizures. Epilepsy can present as heterogenous set of clinical symptoms and is related to extremely varied etiologies. Some epilepsies are triggered by antineuronal autoantibodies and/or complicated by a status epilepticus. These conditions may induce brain atrophy, and severe neurological sequels.

The severity of these epilepsies requires significant efforts to (i) identify new therapeutic strategies able to control the evolution of dysimmune encephalitis and refractory status epilepticus, (ii) to identify their etiologies and (iii) to propose neuroprotective strategies.

Therefore, the investigators will organize a collection of biological samples (blood, cerebrospinal fluid, post-mortem brain tissues) and paraclinical data (electroencephalogram, evoked potential, CT, MRI) in patients with severe epilepsies, whether or not associated with autoantibodies, and/or evolving into status epilepticus.

This study should bring new insights allowing to better understand mechanisms that trigger the emergence of an epileptic brain (epileptogenesis) through :

(i) the identification and characterization of new pathophysiological pathways involving autoimmunity directed against the cerebral cortex and associated with severe epilepsy (ii) the identification and characterization of pathophysiological pathways participating in the excitotoxicity observed in status epilepticus.

ELIGIBILITY:
Inclusion Criteria:

Group 1:

* Patients aged 2 years or above, with status epilepticus.
* Affiliation to a French social security system excluding "Aide Médicale" Etat (AME).
* Patients or relatives have been informed and given free informed and written consent to participate
* Patients under legal protection (guardianship, curatorship) or not

Group 2:

* Patients aged 2 years or above, with clinical signs of epilepsy associated to dysimmune encephalitis.
* Affiliation to a French social security system excluding "Aide Médicale" Etat (AME).
* Patients or relatives have been informed and given free informed and written consent to participate
* Patients under legal protection (guardianship, curatorship) or not

Group 3:

* Patients aged 18 years or above, without status epilepticus and/or dysimmune encephalitis.
* Affiliation to a French social security system excluding "Aide Médicale" Etat (AME).
* Patients or relatives have been informed and given free informed and written consent to participate
* Patients under legal protection (guardianship, curatorship) or not

Exclusion Criteria:

Group 1:

* Women with known or clinically detected pregnancy.
* Patient deprived of liberty
* Patients with known neurodegenerative disease.

Group 2:

* Women with known or clinically detected pregnancy.
* Patient deprived of liberty
* Patients have been already treated by corticoids or IgIV.

Group 3:

* Women with known or clinically detected pregnancy.
* Patient deprived of liberty.
* Patients with status epilepticus.
* Patients with known neurodegenerative disease, brain tumor, severe head trauma, meningitis, subarachnoid hemorrhages, stroke.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2020-11-25 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Identification of (i) antibodies in the plasma and in the cerebrospinal fluid of patients with dysimmune encephalitis and (ii) biomarkers for neuronal death in the plasma and in the cerebrospinal fluid of patients with status epilepticus | 9 months
  Looking for antibodies with cell-based binding assay or monospecific recombinant assay. Identification of biomarkers for neuronal death with electrochemiluminometric sandwich immunoassays (Kryptor and ModularE170, Roche Diagnostic)

SECONDARY OUTCOMES:
Identification of new dysimmune abnormalities | 9 months
  Lymphocyte phenotyping, cytokines quantification
Identification of specific EEG patterns associated to dysimmune encephalitis and/or status epilepticus | 9 months
  EEG signals will be reviewed and classifiyed according to a EEG-based seizure build-up score in status epilepticus (EaSiBUSSEs)
Identification of new genetic pathways associated to dysimmune encephalitis and status | 9 months
  Genetic biomarkers
Identification of new metabolic pathway that may participate in the excitotoxicity observed in status epilepticus or dysimmune encephalitis | 9 months
  Looking for diagnostic and prognosis biomarkers. Characterization of the brain cholesterol homeostasis with UPLC-MS/MS method and enzymatic assays. Evaluation of new biomarkers (proteins, lipids, genes).

CONTACTS AND LOCATIONS:
Overall Officials: Vincent NAVARRO, Pr, Principal Investigator — Hôpital Pitié Salpêtrière - Assitance Publique Hôpitaux de Paris
Locations (1):
- Hôpital de la Pitié Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients. Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.